CLINICAL TRIAL: NCT06906536
Title: Examining the Effect of Acute Intermittent Hypoxia on Serum Blood Proteins, Corticospinal Excitability, and Force Control in Persons With Incomplete Spinal Cord Injury
Brief Title: Examining the Effect of Acute Intermittent Hypoxia on Serum Blood Proteins and Lower Limb Function
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Andrew Quesada Tan, Assistant Professor, University of Colorado, Boulder
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23-1275; 1R03HD115657-01 (NIH)
Record Dates: First submitted 2025-03-11; First posted 2025-04-02 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: INCOMPLETE SPINAL CORD INJURY (ASIA D); Able Bodied
Keywords: Acute Intermittent Hypoxia; Spinal cord injury; Force steadiness
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AIH Group (Experimental): Participants will be exposed to 4 consecutive days of acute intermittent hypoxia (AIH): 15, 1.5 min episodes at 9% O2 alternating with 21% O2 at 1 min intervals.
  Interventions: Other: Acute Intermittent Hypoxia (AIH)
- SHAM Group (No Intervention): Participants will be exposed to 4 consecutive days of normoxia: 15, 1.5 min episodes at 21% O2 alternating with 21% O2 at 1 min intervals.

INTERVENTIONS:
Other: Acute Intermittent Hypoxia (AIH) — 4 consecutive days of 15, 1.5 min episodes at 9% O2 (AIH) alternating with 21% O2 at 1 min intervals
  Arms: AIH Group

SUMMARY:
The goal of this study is to clarify mechanisms of acute intermittent hypoxia and to examine the effect on lower limb function in persons with chronic, incomplete spinal cord injury.

DETAILED DESCRIPTION:
The goal of this study is to clarify mechanisms of acute intermittent hypoxia by examining changes in blood biomarkers, neural excitability, and hemoglobin mass. We also aim to clarify how these changes relate to changes in lower limb function in persons with chronic, incomplete spinal cord injury by measuring force steadiness and voluntary muscle activation.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years old (the latter to reduce likelihood of heart disease)
* Medically stable with medical clearance from physician to participate
* Motor-incomplete spinal cord injuries at or below C2 and at or above L5
* AIS A-D at initial screen, or other non-traumatic spinal cord injury disorders (e.g. multiple sclerosis, ALS, tumors, acute transverse myelitis, etc.)
* More than 1 year since iSCI to minimize confounds of spontaneous neurological recovery
* Ability to advance one step overground with or without assistive devices;

Exclusion Criteria:

* Severe concurrent illness or pain
* Recurrent autonomic dysreflexia
* History of cardiovascular/pulmonary complications
* Concurrent physical therapy
* Pregnant at time of enrollment or planning to become pregnant
* Untreated painful musculoskeletal dysfunction, fracture or pressure sore
* History of seizures or epilepsy
* Recurring headaches
* Concussion within the last six months
* Depression or manic disorder
* Metal implants in the head, or pacemaker
* Aversion to needles

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change in Serum Blood Brain Derived Neurotrophic Factor | Baseline, Day 1, Day 3, and Day 4
  Serum blood brain derived neurotrophic factor (pg/mL) will be assessed using enzyme-linked immunosorbent assay. Blood will be sampled prior to AIH and within 1 hour following the 1st, 3rd, and 4th AIH exposure.
Change in Serum Serotonin | Baseline, Day 1, Day 3, and Day 4
  Serum serotonin (ng/mL) be assessed using enzyme-linked immunosorbent assay. Blood will be sampled prior to AIH and within 1 hour following the 1st, 3rd, and 4th AIH exposure.
Change in the Transcranial Magnetic Stimulation Recruitment Curve Slope | Baseline and Day 4
  The mean motor evoked potential response will be plotted against the corresponding stimulation intensity (% resting motor threshold) to produce a stimulus-response curve at 20% and 40% of maximum. We will measure TMS before the start of 4 consecutive days of AIH exposure. We will measure TMS within 24 hours of the final AIH exposure.
Change in Force Steadiness | Baseline and Day 4
  The coefficient of variation of force will be calculated in both plantarflexion and dorsiflexion at 20% and 40% of maximum. We will measure coefficient of variation of force before the start of 4 consecutive days of AIH exposure. We will measure coefficient of variation of force within 24 hours of the final AIH exposure.
Change in Central Activation Ratio | Baseline and Day 4
  We will measure the central activation ratio using supramaximal electrical stimulus over a peripheral nerve during maximum voluntary activation. We will measure the central activation ratio before the start of 4 consecutive days of AIH exposure. We will measure the central activation ratio within 24 hours of the final AIH exposure.
Change in hemoglobin mass | Baseline and Day 4
  Using the optimized carbon monoxide rebreathing procedure we will evaluate hemoglobin concentration, carboxyhemoglobin, and hematocrit to calculate total hemoglobin mass, blood volume, and plasma volume. The optimized carbon monoxide rebreathing procedure will be done prior to the first hypoxia exposure and following the 4th hypoxia exposure.
Change in Serum Erythropoetin | Baseline, Day 1, Day 3, and Day 4
  Serum erythropoetin (mU/mL) will be assessed using enzyme-linked immunosorbent assay. Blood will be sampled prior to AIH and within 1 hour following the 1st, 3rd, and 4th AIH exposure.

SECONDARY OUTCOMES:
Axial damage ratio | Baseline
  Using MRI, we will quantify the axial damage ratio. Prior to participation in the study we will obtain an MRI for quantification of axial damage ratio
6-Minute Walk Test | Baseline and Day 4
  We will assess the distance walked in 6-minutes. The 6-minute walk test will be completed prior to the first exposure to hypoxia and following the 4th exposure of hypoxia.
10-Meter Walk Test | Baseline and Day 4
  We will assess how long it takes subjects to walk 10 meters. The 10-Meter walk test will be done prior to the first hypoxia exposure, and following the 4th hypoxia exposure.

CONTACTS AND LOCATIONS:
Locations (1):
- Andrew Tan, Boulder, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided